CLINICAL TRIAL: NCT03141567
Title: LYmphangiogenesis FacTors in Heart Failure States (LYFT-HF Study)
Brief Title: LYmphangiogenesis FacTors in Heart Failure States
Acronym: LYFT-HF
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00062457
Record Dates: First submitted 2017-04-27; First posted 2017-05-05 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Normal Ejection Fraction
Keywords: Lymphangiogenesis; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — plasma or serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Outpatient: Individuals undergoing clinically indicated Right Heart Catheterization.
- Inpatient: Individuals undergoing clinically indicated Right Heart Catheterization.

SUMMARY:
Heart failure often causes fluid to accumulate in the body, leading to congestion and swelling. However, some people who have had heart failure for a long time seem to have very little congestion or swelling, even when the heart failure is poorly treated. The investigators think that this is because lymphatic vessels are able to grow and remove fluid to prevent congestion. The investigators do not know how lymphatic vessels grow. This study will investigate the blood levels of various proteins to try to figure out how the lymph vessels of people with long-standing heart failure might grow.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing clinically indicated right heart catheterization.

Exclusion Criteria:

* Unable to provide consent.
* Use of medications which may alter lymphangiogenesis factor expression within 365 days
* Thalidomide, lenalidomide, pomalidomide
* Bevacizumab
* Any cytotoxic chemotherapy agents
* Pregnant
* Any potentially pregnant patient (based on age and gender) undergoes Beta Human chorionic gonadotropin testing as standard of care prior to any right heart catheterization.
* Active cancer within 365 days
* Diagnosis of familial or secondary lymphedema
* Treatment of active bacterial infection within 7 days
* Active inflammatory rheumatologic disease requiring anti-inflammatory therapy administration within 60 days
* Conditions
* Systemic lupus erythematosus
* Rheumatoid arthritis
* Scleroderma
* Inflammatory myositis
* Vasculitis
* Behcet's disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Inpatient and Outpatient individuals undergoing clincially-indicated right heart catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Vascular Endothelial Growth Factor (VEGF) Levels | At time of right heart catheterization
  VEGF levels in systemic venous, pulmonary arterial, and pulmonary venous samples in participants with left heart failure versus those without left heart failure.

SECONDARY OUTCOMES:
Lymphangiogenesis factors and Pulmonary Capillary Wedge Pressure (PCWP) | At time of right heart catheterization
  Correlation between above lymphangiogenesis factors and pulmonary capillary wedge pressure, right atrial pressure, and cardiac output gathered from right heart catheterization.
Lymphangiogenesis and Heart failure severity | At time of right heart catheterization
  Correlation between lymphangiogenesis factors and heart failure symptom severity as determined by the Kansas City Cardiomyopathy Questionnaire
Lymphangiogenesis and 6 minute hall walk | At time of right heart catheterization
  Correlation between lymphangiogenesis factors and 6 minute walk distance.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Houston, M.D., Principal Investigator — Assistant Professor
Locations (2):
- United States (2):
  - Ralph H. Johnson VAMC, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No